CLINICAL TRIAL: NCT01223313
Title: A Multicenter, Open-Label, Non-Comparative Study of the Safety and Contraceptive Efficacy of the Woman's Condom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCN008
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Contraception
Keywords: Contraception; Woman's Condom; Female Condom; Condom

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Woman's Condom (Experimental): The Woman's Condom (WC) is an investigational device manufactured by Shanghai Dahua Medical Apparatus Corp., Ltd (Dahua). Dahua's quality management system complies with ISO9001:2000, ISO13485:2003, MDD93/42/EEC. The WC consists of a 0.03-mm-thick pliable plastic pouch that easily conforms to the shape of the vagina. It is 22.9 cm (± 0.3 cm)(9 inches ± 0.1 inch) long and has a flexible soft outer ring that is designed to hug the external genitalia. The foam shapes on the outside of the pouch cling lightly to vaginal walls, ensuring stability of the device. The insertion capsule is made from dissolvable polyvinyl alcohol (PVA) and is similar to the PVA used in C-Film (Apothecus Pharmaceutical Corporation, New York, NY). The WC is a non-lubricated device. It is supplied with water-soluble lubricant with a chemical composition similar to a commercially available lubricant used in previous studies of the WC. Women will receive instruction sheets on the use of the WC and lubricant.
  Interventions: Device: Woman's Condom

INTERVENTIONS:
Device: Woman's Condom — The Woman's Condom (WC) is an investigational device manufactured by Shanghai Dahua Medical Apparatus Corp., Ltd (Dahua). Dahua's quality management system complies with ISO9001:2000, ISO13485:2003, MDD93/42/EEC. The WC consists of a 0.03-mm-thick pliable plastic pouch that easily conforms to the shape of the vagina. It is 22.9 cm (± 0.3 cm)(9 inches ± 0.1 inch) long and has a flexible soft outer ring that is designed to hug the external genitalia. The foam shapes on the outside of the pouch cling lightly to vaginal walls, ensuring stability of the device. The insertion capsule is made from dissolvable polyvinyl alcohol (PVA) and is similar to the PVA used in C-Film (Apothecus Pharmaceutical Corporation, New York, NY). The WC is a non-lubricated device. It is supplied with water-soluble lubricant with a chemical composition similar to a commercially available lubricant used in previous studies of the WC. Women will receive instruction sheets on the use of the WC and lubricant.

SUMMARY:
WHAT IS THE FEMALE CONDOM? The female condom being examined in this study is investigational (experimental) and is not yet approved by the Food and Drug Administration (FDA). The female condom is made up of a pouch that adjusts to the shape of the vagina. The female condom that will be used in this study is not lubricated, but a water-based lubricant will be provided for you to use with it. Also, the female condoms used in this study will be provided to you at no cost.

WHY IS THIS STUDY BEING DONE?

The purpose of this study is to find out:

* How well the female condom works to prevent pregnancy
* How well the female condom works to prevent transmission of sexually transmitted diseases
* How safe the female condom is to use
* If urinary tract infections and symptomatic vaginal infections occur while using the female condom
* How well women like the female condom
* How well the female condom performs.

WHAT DOES THE STUDY INVOLVE? There will be approximately 10 clinics in the study with about 500 women from all over the United States participating in this study. You are being asked to participate in a research study because you are a woman between the ages of 18 and 40, are in general good health, have regular menstrual cycles, do not want to become pregnant for at least the next 7 months, and are willing to rely on the female condom as your primary method of contraception during study participation.

HOW LONG DOES THE STUDY LAST? Enrollment for this study is expected to last about 12 months. You will need to come to the clinic for a screening/admission visit and then 2 or more visits. You will also be asked to complete a diary every day about your use of the female condoms. The clinical staff will help set up your planned clinical visits during the study.

DETAILED DESCRIPTION:
This is a Phase III multicenter, open-label, non-comparative trial of the Woman's Condom to evaluate contraceptive efficacy as the primary method of contraception. Secondary evaluations include safety assessment, incidence of UTIs, symptomatic vaginal infection, performance of the Woman's Condom (clinical breakage, slippage, misdirection, and invagination) and overall acceptability of the product. We will perform a Substudy to assess the semen biomarker as a means of detecting product failure in a subset of subjects.

ELIGIBILITY:
Inclusion Criteria

To enroll into the clinical trial, potential subjects must:

1. Be healthy women, who are sexually active, at risk for pregnancy and desiring contraception.
2. Be within the age range of 18 through 40 years inclusive at enrollment.
3. Have a negative urine pregnancy test at the admission visit.
4. Have a history of regular cyclic menses with a usual length of 21 to 35 days when not using hormonal contraception.
5. Have one menses after switching from oral contraceptives to using the Woman's Condom.
6. Have at least one spontaneous menstrual cycle (two menses) following a pregnancy that ended at 14 or more weeks gestation.
7. Have at least one cycle (two menses) after an abortion at less than 14 weeks gestation.
8. Be willing to accept a risk of pregnancy.
9. Be willing to engage in at least four acts of heterosexual vaginal intercourse per month for a period of 6 months.
10. Be willing to only use the study product as the primary method of contraception over the course of the study.
11. Be capable of using the study product properly and agree to observe all study directions and requirements.
12. Be willing to keep a diary to record coital information, product use information, information about the use of other vaginal products, and any symptoms, which occurred in her or her partner over the course of study participation.
13. Be willing to state that, to her best knowledge, her sexual partner(s):

    1. Has not had a vasectomy or been previously diagnosed as infertile.
    2. Has not been previously diagnosed or suspected of HIV unless he has subsequently had a negative HIV test.
    3. Has not been known to have engaged in homosexual intercourse in the past 5 years unless he has had negative HIV test results since then.
    4. Has not shared injection drug needles in the past unless he has had a negative HIV test at least 6 weeks since last use.
    5. Has no known history of allergy or sensitivity to polyurethane (condom pouch), polyvinyl alcohol (capsule), or other water-based lubricants such as Astroglide.
14. Agree not to participate in any other clinical trials during the course of this study.
15. Be willing to give written informed consent to participate in the trial.

Exclusion Criteria

To enroll into the clinical trial, potential subjects must not:

1. Have a history of allergy or sensitivity to polyurethane (condom pouch), polyvinyl alcohol (capsule), or other water-based lubricants such as Astroglide.
2. Have current UTI or symptomatic vaginal infection as confirmed by dipstick urinalysis, or if needed by a urine culture or wet mount (see Schedule of Assessments for definitions), unless treated and proof of cure is documented by a negative test result performed at least 2 weeks post-treatment.
3. Have evidence of Chlamydia trachomatis or Neisseria gonorrhea infection unless she and her partner(s) complete treatment and proof of cure is documented for the subject only by a negative test result performed at least 3 weeks post-treatment.
4. Be pregnant, have a suspected pregnancy or desire to become pregnant during the course of the study.
5. Have a history of infertility or pelvic inflammatory disease without a subsequent spontaneous intrauterine pregnancy.
6. Have been diagnosed with pelvic inflammatory disease (PID) without a subsequent intrauterine pregnancy.
7. Be in a monogamous relationship of less than 4 months with their partner.
8. Have any contraindications to pregnancy (medical condition) or regularly use category D or X or exclusionary medications listed in Appendix F.
9. Have shared injection drug needles in the past unless has a negative HIV test at least 6 weeks since last use.
10. Have known or suspected to have an HIV infection.
11. Have been diagnosed with genital herpes simplex virus (HSV), with the first occurrence (initial episode) within 3 months prior to screening or have clinical evidence of HSV on exam.
12. Be lactating or breastfeeding.
13. Have any clinically significant abnormal vaginal bleeding or spotting within the month prior to screening.
14. Have had vaginal or cervical biopsy or vaginal surgery within 3 months prior to screening.
15. Have used vaginal or systemic antibiotics or antifungal agents within 14 days prior to screening or enrollment.
16. Have received a Depo-Provera® injection in the 9 months prior to enrollment (this exclusionary time period can be shortened to 6 months if the subject has also had 2 spontaneous menstrual cycles [requires minimum of 3 menses] that meet criteria for normal menstrual cycles).
17. Have an abnormal Pap test based on the following criteria:

    * Pap test in the past 15 months with ASC-US unless:

      * less than 21 years of age;
      * a repeat Pap test at least 6 months later was normal;
      * reflex HPV testing was performed and was negative for high-risk HPV; or
      * a colposcopy (with or without biopsy) found no evidence of dysplasia requiring treatment or treatment was performed and follow-up at least 6 months after the treatment showed no evidence of disease;
    * Pap test in the past 15 months with LSIL unless:

      * less than 21 years of age;
      * a colposcopy (with or without biopsy) found no evidence of dysplasia requiring treatment or treatment was performed and follow-up at least 6 months after the treatment showed no evidence of disease;
    * Pap test in the past 15 months with ASC-H, atypical glandular cells, or HSIL unless colposcopy and/or treatment was performed and follow-up at least 6 months after the colposcopy and/or treatment showed no evidence of disease;
    * Pap test in the past 15 months with malignant cells.
18. Have a past (within 12 months) or current history of alcohol or drug [recreational, prescription or over-the-counter (OTC)] abuse.
19. Have taken an investigational drug or used an investigational device within the past 30 days.
20. Have previously participated in or completed this study.
21. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study. For example, if the subject is found to have Condyloma Accuminata, the investigator can decide whether to exclude the subject or not, depending on its location and if use of the condom may be painful for the subject.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 511 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - California Family Health Council, Inc, Los Angeles, California
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - NYU Medical Center Family Planning, New York, New York
  - Columbia University, New York, New York
  - University of Cininnati College of Medicine, Cincinnati, Ohio
  - Oregon Health Scieces University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center Dept. of OB/Gyn, Dallas, Texas
  - Jones Institute of Reproductive Medicine, Norfolk, Virginia

REFERENCES:
- [Derived] Walsh TL, Snead MC, St Claire BJ, Schwartz JL, Mauck CK, Frezieres RG, Blithe DL, Archer DF, Barnhart KT, Jensen JT, Nelson AL, Thomas MA, Wan LS, Weaver MA. Comparison of self-reported female condom failure and biomarker-confirmed semen exposure. Contraception. 2019 Nov;100(5):406-412. doi: 10.1016/j.contraception.2019.07.143. Epub 2019 Aug 2. PMID 31381878
- [Derived] Chen BA, Blithe DL, Muraguri GR, Lance AA, Carr BR, Jensen JT, Kimble TD, Murthy AS, Schreiber CA, Thomas MA, Walsh TL, Westhoff C, Burke AE. Acceptability of the Woman's Condom in a phase III multicenter open-label study. Contraception. 2019 Jun;99(6):357-362. doi: 10.1016/j.contraception.2019.02.006. Epub 2019 Mar 6. PMID 30849305

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was designed to enroll 500 participants. However, the study enrolled 511 participants.
Groups:
- Woman's Condom: The Woman's Condom (WC) is an investigational device manufactured by Shanghai Dahua Medical Apparatus Corp., Ltd (Dahua). The WC consists of a 0.03-mm-thick pliable plastic pouch that easily conforms to the shape of the vagina. It is 22.9 cm (± 0.3 cm)(9 inches ± 0.1 inch) long and has a flexible soft outer ring that is designed to hug the external genitalia. The insertion capsule is made from dissolvable polyvinyl alcohol (PVA) and is similar to the PVA used in C-Film (Apothecus Pharmaceutical Corporation, New York, NY). The WC is a non-lubricated device. It is supplied with water-soluble lubricant with a chemical composition similar to a commercially available lubricant used in previous studies of the WC.
Period: Overall Study
Arm/Group | Woman's Condom
Started | 511
Completed | 278
Not Completed | 233

BASELINE CHARACTERISTICS:
Arm/Group | Woman's Condom
Number analyzed (Participants) | 511
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 511
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 511
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 511

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Pregnancy Probabilities With Typical Use
Description: Kaplan-Meier methods will be used to estimate the six-month cumulative pregnancy probability of women in the MITT population. Pregnancies are not included if they are found to have occurred before a subject was enrolled or after she has discontinued using the study product as her primary method of contraception. The pregnancy probability is reported as a percentage.
Time Frame: Assessed at 1 Month, 3 Months, and 6 Months, up to 6 Months
Population: enrolled subjects whose diaries indicated they had at least one episode of coitus while using the assigned study product and for whom there is at least one report of pregnancy status.
Measure: Number (95% Confidence Interval); unit: percentage of probability
Groups:
- Woman's Condom: The Woman's Condom (WC) is an investigational device manufactured by Shanghai Dahua Medical Apparatus Corp., Ltd (Dahua). Dahua's quality management system complies with ISO9001:2000, ISO13485:2003, MDD93/42/EEC. The WC consists of a 0.03-mm-thick pliable plastic pouch that easily conforms to the shape of the vagina. It is 22.9 cm (± 0.3 cm)(9 inches ± 0.1 inch) long and has a flexible soft outer ring that is designed to hug the external genitalia. The foam shapes on the outside of the pouch cling lightly to vaginal walls, ensuring stability of the device. The insertion capsule is made from dissolvable polyvinyl alcohol (PVA) and is similar to the PVA used in C-Film (Apothecus Pharmaceutical Corporation, New York, NY). The WC is a non-lubricated device. It is supplied with water-soluble lubricant with a chemical composition similar to a commercially available lubricant used in previous studies of the WC.
Arm/Group | Woman's Condom
Number analyzed (Participants) | 401
percentage of probability
  1 Month Pregnancy Probability | 0.5 [0.0 to 1.2]
  3 Month Pregnancy Probability | 1.4 [0.1 to 2.6]
  6 Month Pregnancy Probability | 4.0 [1.6 to 6.3]

2. Secondary Outcome: 6 Month Pregnancy Probabilities With Perfect Use
Description: Kaplan-Meier methods will be used to estimate the six-month cumulative pregnancy probability of women in the Efficacy Evaluable population. Each woman in the Efficacy Evaluable population contributes efficacy for menstrual cycles where she has used the assigned product consistently and correctly as reflected in her diary recordings. Pregnancies that are found to have occurred before a subject was enrolled or after she has discontinued using the study product as her primary method of contraception are not included. The pregnancy probability is reported as a percentage.
Time Frame: Assessed at 1 Month, 3 Months, and 6 Months, up to 6 Months
Population: enrolled subjects whose diaries indicated they had used the assigned study product correctly for every coital act for at least one menstrual cycle and for whom there is at least one report of pregnancy status.
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Woman's Condom
Number analyzed (Participants) | 277
percentage of probability
  1 Month Pregnancy Probability | 0.0 [0.0 to 0.0]
  3 Month Pregnancy Probability | 0.4 [0.0 to 1.1]
  6 Month Pregnancy Probability | 2.6 [0.4 to 4.7]

3. Secondary Outcome: Incidence of Chlamydia During the Study
Description: Incidence of acquisition of Chlamydia evaluated at screening and end of the study.
Time Frame: Visit 1 (Screening) and Visit 3 (Exit), up to 6 months
Population: Subjects that used at least one Woman's Condom and had chlamydia test performed at the respective visits
Measure: Count of Participants; unit: Participants
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
Participants
  Positive Chlamydia at Visit 1/Screening: number analyzed (Participants) | 394
  Positive Chlamydia at Visit 1/Screening | 7
  Positive Chlamydia at Visit 3/Exit: number analyzed (Participants) | 368
  Positive Chlamydia at Visit 3/Exit | 4

4. Secondary Outcome: Incidence of Gonorrhea During the Study
Description: Incidence of acquisition of Gonorrhea evaluated at screening and end of the study.
Time Frame: Visit 1 (Screening) and Visit 3 (Exit), up to 6 months
Population: Subjects that used at least one Woman's Condom and had gonorrhea test performed at the respective visits
Measure: Count of Participants; unit: Participants
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
Participants
  Positive Gonorrhea at Visit 1/Screening: number analyzed (Participants) | 394
  Positive Gonorrhea at Visit 1/Screening | 4
  Positive Gonorrhea at Visit 3/Exit: number analyzed (Participants) | 368
  Positive Gonorrhea at Visit 3/Exit | 6

5. Secondary Outcome: Change From Baseline in Urinary Tract Infections (UTIs)
Description: Change from Baseline of urinary tract infections (UTIs)
Time Frame: Visit 1/Screening and Visit 3/Exit, up to 6 months
Population: only subjects that had both a baseline and exit visit UTI screening were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Woman's Condom
Number analyzed (Participants) | 378
Participants
  Subjects with No Change from Baseline | 373
  Subjects Improved from Baseline | 2
  Subjects Worsened from Baseline | 3

6. Secondary Outcome: Change From Baseline in Bacterial Vaginosis (BV)
Description: Change from Baseline of bacterial vaginosis (BV)
Time Frame: Visit 1/Screening and Visit 3/Exit, up to 6 months
Population: only subjects that had both a baseline and exit visit BV screening were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Woman's Condom
Number analyzed (Participants) | 234
Participants
  Subjects with No Change from Baseline | 222
  Subjects Improved from Baseline | 3
  Subjects Worsened from Baseline | 9

7. Secondary Outcome: Change From Baseline in Monilia
Description: Change from Baseline of Monilia
Time Frame: Visit 1/Screening and Visit 3/Exit, up to 6 months
Population: only subjects that had both a baseline and exit visit monilia screening were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Woman's Condom
Number analyzed (Participants) | 10
Participants
  Subjects with No Change from Baseline | 10
  Subjects Improved from Baseline | 0
  Subjects Worsened from Baseline | 0

8. Primary Outcome: 6 Month Pearl Rate With Typical Use
Description: Pearl rate will be calculated based on the number of woman-months that the subject was at risk for pregnancy. Woman-months of pregnancy risk is defined as the (last date study product considered primary means of contraception - date of enrollment + 1) / 30.4 for women who are not pregnant and as (date of conception - date of enrollment + 1) / 30.4 for women who became pregnant during the study.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Number; unit: Pregnancies per 100 women-years
Units Other Than Participants: Months
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
Number analyzed (Months) | 2241
Pregnancies per 100 women-years | 8.03

9. Secondary Outcome: Incidence of Trichomoniasis During the Study
Description: Incidence of acquisition of Trichomoniasis evaluated at screening and end of the study.
Time Frame: Visit 1 (Screening) and Visit 3 (Exit), up to 6 months
Population: Subjects that used at least one Woman's Condom and had trichomoniasis test performed at the respective visits. Subjects were only tested for trichomoniasis if clinically indicated. Therefore, not all subjects were tested. Only 12 subjects were tested for trichomoniasis based on clinical indication for testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Woman's Condom
Number analyzed (Participants) | 12
Participants
  Positive Gonorrhea at Visit 1/Screening | 3
  Positive Gonorrhea at Visit 3/Exit | 0

10. Secondary Outcome: Number of Women That Preferred Female Condom Over Male Condom After Cycle 6
Description: Acceptability of the Woman's Condom as measured by an acceptability questionnaire administered at study exit (visit 3, after menstrual cycle 6 or early discontinuation).
Time Frame: Visit 3 (Cycle 6), up to 6 months
Population: Subjects that completed the questionnaire at exit visit were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Woman's Condom
Number analyzed (Participants) | 337
Participants | 81

11. Secondary Outcome: Percentage of Uses With Clinical Breakage With the Woman's Condom
Description: Performance of the Woman's Condom as assessed by self-reported clinical breakage based on percent of uses. Breakage of the female condom during intercourse or during withdrawal of the condom from the vagina. Clinical breakage is breakage with potential adverse health consequences and includes events in which the outer frame or ring breaks. It is calculated by dividing the number of female condoms reported to have broken during intercourse or withdrawal by the number of female condoms used during intercourse.
Time Frame: Up to 6 months of use
Population: Subjects that used the Woman's Condom were analyzed
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
percentage | 1.2 (6.44)

12. Secondary Outcome: Percentage of Uses With Misdirection With the Woman's Condom
Description: Performance of the Woman's Condom as assessed by self-reported misdirection based on percent of uses. Vaginal penetration whereby the penis is inserted between the female condom and the vaginal wall and is calculated by dividing the number of reported incidences of misdirection by the number of female condoms used during intercourse.
Time Frame: Up to 6 months of use
Population: Subjects that used the Woman's Condom were analyzed
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
percentage | 2.2 (7.79)

13. Secondary Outcome: Percentage of Uses With Slippage With the Woman's Condom
Description: Performance of the Woman's Condom as assessed by self-reported slippage based on percent of uses. A female condom that slips completely out of the vagina during intercourse and is calculated by dividing the number of female condoms that slipped during intercourse by the number of female condoms used during intercourse.
Time Frame: Up to 6 months of use
Population: Subjects that used the Woman's Condom were analyzed
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
percentage | 4.3 (13.24)

14. Secondary Outcome: Percentage of Uses With Invagination With the Woman's Condom
Description: Performance of the Woman's Condom as assessed by self-reported invagination based on percent of uses. As part of the entire external component of the female condom being pushed into the vagina during intercourse and is calculated by dividing the number of reported incidences of invagination during intercourse by the number of female condoms used during intercourse.
Time Frame: Up to 6 months of use
Population: Subjects that used the Woman's Condom were analyzed
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
percentage | 1.9 (7.48)

15. Secondary Outcome: Percentage of Uses With Total Clinical Failure With the Woman's Condom
Description: Performance of the Woman's Condom as assessed by total clinical failure based on percent of uses. Total Clinical Failure is defined as the number of female condoms that clinically break, slip, or are associated with reported incidences of misdirection or invagination during intercourse (i.e., any event that might lead to semen spillage) and is calculated by dividing the sum of these events by the number of female condoms used during intercourse.
Time Frame: Up to 6 months of use
Population: Subjects that used the Woman's Condom were analyzed
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Woman's Condom
Number analyzed (Participants) | 405
percentage | 8.0 (16.31)

ADVERSE EVENTS:
Time Frame: 6 months, immediately after informed consent has been obtained and lasts through the study Exit Visit, up to 6 months.
Description: For this study, an Adverse Event (AE) is defined as one following: 1) any genital or urinary tract problem that lasts more than an hour, 2) any non-genital/urinary tract problem that is at least possibly related to condom use, or 3) a serious adverse event. The transient symptoms associated with the use of the study condom will not be reported as AEs. Those symptoms include irritation, itching, burning, rash, abnormal discharge (not including gel), odor, or pain or difficulty in urination.
Arm/Group | Woman's Condom
All-Cause Mortality (participants affected / at risk) | 0/405
Serious Adverse Events (participants affected / at risk) | 1/405
Other Adverse Events (participants affected / at risk) | 102/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Woman's Condom (N=405)
Convulsion (Nervous system disorders) | 1 (1) — Hospitalized for seizure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Woman's Condom (N=405)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Cervicitis trichomonal (Infections and infestations) | 1 (1)
Chlamydial infection (Infections and infestations) | 6 (6)
Fungal infection (Infections and infestations) | 2 (2)
Gonorrhoea (Infections and infestations) | 2 (2)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 17 (17)
Vaginitis bacterial (Infections and infestations) | 19 (19)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 17 (17)
Smear cervix abnormal (Investigations) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 6 (6)
Micturition urgency (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 4 (4)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 2 (2)
Genital pain (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 6 (6)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 7 (7)
Vaginal disorder (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Vaginal odour (Reproductive system and breast disorders) | 5 (5)
Vaginal swelling (Reproductive system and breast disorders) | 1 (1)
Vulval disorder (Reproductive system and breast disorders) | 2 (2)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 7 (7)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 19 (19)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes